CLINICAL TRIAL: NCT00791583
Title: Emergency Medicine Residents Performance in Maximum Barrier Precautions During Central Venous Catheter Placement: Effect of Stimulation-based Training
Brief Title: ED Residents MBP During CVC Placement: Sim Lab Based Training
Acronym: EM CVC MBP
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Principal Investigator, Hassan Khouli, MD, St. Luke's-Roosevelt Hospital Center
Other Study IDs: 08-007
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Nosocomial Infections
Keywords: Emergency Medicine (EM); Central Venous Catheter (CVC); Maximal Barrier Precaution (MBP); Precaution Technique during Central Venous Cathether Placement
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Baseline performance in maximal barrier precaution technique of Emergency Medicine (EM) residents, certified in CVC placement, is poor
2. Simulation-based training in maximal barrier precaution technique during central venous catheter (CVC) placement will improve baseline performance of EM residents

DETAILED DESCRIPTION:
Central line associated bloodstream infection (CL-ABI) is an important and preventable cause of nosocomial infections and is responsible for considerable morbidity and mortality. It is estimated that 5 to 26% of patients experience an infectious complication from their central venous catheter [1]. In the United States, it is estimated that nearly 50,000 patients develop central line associated bloodstream infections in the ICUs annually, at a rate of approximately 5 infections per 1000 catheter days [2] and as many as 15,000 deaths annually. Central line associated bloodstream infections are also associated with increased hospital and ICU lengths of stay in the ICU (2). Estimates of the cost of CL-ABI to hospitals range from $25,000 to $65,000 per patient [3, 4].

The Centers for Disease Control have published guidelines for the prevention of CL-ABI that represent a collaborative effort by a multidisciplinary coalition of professional organizations that provide evidence based recommendations to prevent catheter related infections [5]. The interventions emphasize five distinct practices, including: education and training of healthcare providers who place and care for catheters, utilizing maximum sterile barrier precautions during catheter placement, skin preparation using 2% chlorhexidine, avoiding routine replacement of central lines as a strategy to reduce infection, and using antiseptic or antibiotic coated lines in the event that infection rates remain high despite adherence to the above measures [5].

Several studies have demonstrated impressive reductions in CL-ABI from the application of these strategies, ranging from 18 to 100% reductions and realizing significant reductions in mortality and cost [2]. The simple introduction of maximum sterile barrier precautions to insert central lines has been observed to dramatically reduce infection rates for over a decade [6]. However, the CDC's guidelines, despite their seeming simplicity, have been found to be frequently insufficiently applied, whether by ignorance or omission [2].

In the past 12 months there have been a total 24 documented central venous line (CVL) infections at SLRHC with cumulative rate of infection of 3.8 per 1000 central line days. These infection rate figures are above the benchmark experience. For SLRHC the cost incurred over the past 12 months is estimated to be $1,080,000.

Training and education of healthcare personnel and the utilization of maximum sterile precautions are two important areas. Residents still most frequently learn central line placement techniques by the "see one, do one, teach one" method, which by its very definition allows for a multitude of techniques in practice. While this teaching theoretically includes the utilization of maximal sterile precautions for central line placement, the focus of teaching, and of residents' anxieties, is most often focused on the proper placement of the line, not the sterile technique used to place it. In emergency medicine, residents also frequently learn procedures in an emergent environment- where attention to maximum sterile precautions may be less than ideal. Guzzo et al found in particular that mentors of trainees performing CVC placements in both emergent and non-emergent situations were significantly less likely to consistently utilize maximum sterile precautions [8]. Furthermore, in a study of a video-based training on sterile technique in CVC insertion in a trauma resuscitation unit that evaluated only non-emergent CVC placements, a total of 5 cases of central- catheter- related bacteremia were reported on just 68 patients, and even with video based training, 26% of residents continued to have infractions in their compliance with sterile precautions [9].

Medical simulators allow residents to practice skills in a realistic and interactive environment that minimizes risk to patients. Studies have found simulation to be an effective means for teaching skills as diverse as ACLS and airway management to laparoscopic surgical skills [10,11,12]. Additionally, the use of audio-visual equipment in a medical simulator to record a resident's performance gives valuable firsthand feedback that is otherwise not available, as it allows residents to visualize their own missteps [13]. This is hypothesized to be of particular value in the proper acquisition of physical skills such as maximum sterile precautions. Furthermore, the Society for Academic Medicine has recently published a consensus paper outlining a research agenda for the use of simulation in Emergency Medicine that identifies procedural training as a priority area and notes that it is "an incompletely tested assessment method for the range of procedural skills required of emergency physicians [14]." The paper goes on to state that:

"Competency" must be defined precisely for every procedure. Each step must be identified, and the proper sequence of those steps must be established. Objective checklists and expert scoring systems must be created, and training and assessment methodologies must be validated. [14] With this in mind, the Department of Emergency Medicine has recently approved a training policy in aseptic technique during central venous access placement (see attached copy). All EM residents will be trained in MBP techniques in the Sim Lab. Training will include baseline assessment of residents skills in maintaining maximum sterile precautions using a standardized scoring tool, videotape training, short exam, and individual simulated debriefing on performance of correct MBP with follow up assessment and training as needed.

We plan to collect data prospectively on all EM residents who will undergo evaluation and training in maximum barrier precaution during CVC placement. Data will be reviewed and analyzed for future research publication

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine (EM) residents who are eligible by their residency training program to place a CVC and will be undergoing evaluation and training in MBP according to their department training policy.

Exclusion Criteria:

* Residents who refuse to have their data collected for the sake of this study and later analyzed for publication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency Medicine Residents
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Emergency Medicine residents' performance in maximal barrier precaution (MBP) technique during central venous catheter (CVC) placement | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Roosevelt Hospital, New York, New York, United States

REFERENCES:
- [Background] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Background] Eggimann P. Prevention of intravascular catheter infection. Curr Opin Infect Dis. 2007 Aug;20(4):360-9. doi: 10.1097/QCO.0b013e32818be72e. PMID 17609594
- [Background] Posa PJ, Harrison D, Vollman KM. Elimination of central line-associated bloodstream infections: application of the evidence. AACN Adv Crit Care. 2006 Oct-Dec;17(4):446-54; quiz 456. doi: 10.4037/15597768-2006-4009. PMID 17091045
- [Background] Shannon RP, Patel B, Cummins D, Shannon AH, Ganguli G, Lu Y. Economics of central line--associated bloodstream infections. Am J Med Qual. 2006 Nov-Dec;21(6 Suppl):7S-16S. doi: 10.1177/1062860606294631. PMID 17077414
- [Background] Bull DA, Neumayer LA, Hunter GC, Sethi GK, McIntyre KE, Bernhard VM, Putnam CW. Improved sterile technique diminishes the incidence of positive line cultures in cardiovascular patients. J Surg Res. 1992 Feb;52(2):106-10. doi: 10.1016/0022-4804(92)90287-a. PMID 1740929
- [Background] Guzzo JL, Seagull FJ, Bochicchio GV, Sisley A, Mackenzie CF, Dutton RP, Scalea T, Xiao Y. Mentors decrease compliance with best sterile practices during central venous catheter placement in the trauma resuscitation unit. Surg Infect (Larchmt). 2006 Feb;7(1):15-20. doi: 10.1089/sur.2006.7.15. PMID 16509781
- [Background] Xiao Y, Seagull FJ, Bochicchio GV, Guzzo JL, Dutton RP, Sisley A, Joshi M, Standiford HC, Hebden JN, Mackenzie CF, Scalea TM. Video-based training increases sterile-technique compliance during central venous catheter insertion. Crit Care Med. 2007 May;35(5):1302-6. doi: 10.1097/01.CCM.0000263457.81998.27. PMID 17414726
- [Background] Wayne DB, Siddall VJ, Butter J, Fudala MJ, Wade LD, Feinglass J, McGaghie WC. A longitudinal study of internal medicine residents' retention of advanced cardiac life support skills. Acad Med. 2006 Oct;81(10 Suppl):S9-S12. doi: 10.1097/00001888-200610001-00004. PMID 17001145
- [Background] Mayo PH, Hackney JE, Mueck JT, Ribaudo V, Schneider RF. Achieving house staff competence in emergency airway management: results of a teaching program using a computerized patient simulator. Crit Care Med. 2004 Dec;32(12):2422-7. doi: 10.1097/01.ccm.0000147768.42813.a2. PMID 15599146
- [Background] Murray D. Clinical simulation: measuring the efficacy of training. Curr Opin Anaesthesiol. 2005 Dec;18(6):645-8. doi: 10.1097/01.aco.0000188419.77140.1a. PMID 16534306
- [Background] Savoldelli GL, Naik VN, Park J, Joo HS, Chow R, Hamstra SJ. Value of debriefing during simulated crisis management: oral versus video-assisted oral feedback. Anesthesiology. 2006 Aug;105(2):279-85. doi: 10.1097/00000542-200608000-00010. PMID 16871061
- [Background] Bond WF, Lammers RL, Spillane LL, Smith-Coggins R, Fernandez R, Reznek MA, Vozenilek JA, Gordon JA; Society for Academic Emergency Medicine Simulation Task Force. The use of simulation in emergency medicine: a research agenda. Acad Emerg Med. 2007 Apr;14(4):353-63. doi: 10.1197/j.aem.2006.11.021. Epub 2007 Feb 15. PMID 17303646
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537